CLINICAL TRIAL: NCT06388564
Title: A Phase 2, Open-Label, Randomized, Multicenter Study to Evaluate the Safety and Efficacy of Axatilimab in Combination With Ruxolitinib in Participants With Newly Diagnosed Chronic Graft-Versus-Host Disease
Brief Title: A Study to Evaluate the Safety and Efficacy of Axatilimab in Combination With Ruxolitinib in Participants With Newly Diagnosed Chronic Graft-Versus-Host Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCA34176-254; 2022-502168-19-00 (Registry Identifier: EU CT Number)
Expanded Access: NCT05544032 (Available)
Record Dates: First submitted 2024-04-25; First posted 2024-04-29 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Chronic Graft-versus-host-disease
Keywords: cGVHD
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — axatilimab; ruxolitinib; Adrenal Cortex Hormones; Prednisone; Prednisolone; Methylprednisolone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment Group A (Experimental): Axatilimab will be administered at a protocol defined starting dose plus ruxolitinib at a protocol defined starting dose.
  Interventions: Drug: Axatilimab; Drug: Ruxolitinib
- Treatment Group B (Experimental): Ruxolitinib will be administered at a protocol defined starting dose.
  Interventions: Drug: Ruxolitinib
- Treatment Group C (Experimental): Corticosteroids alone will be administered at a protocol defined starting dose.
  Interventions: Drug: Corticosteroids

INTERVENTIONS:
Drug: Axatilimab — Axatilimab will be administered at protocol defined dose.
  Arms: Treatment Group A
Drug: Ruxolitinib — Ruxolitinib will be administered at protocol defined dose.
  Arms: Treatment Group A; Treatment Group B
Drug: Corticosteroids — Corticosteroids will be administered at protocol defined dose.
  Other Names: prednisone, prednisolone, methylprednisolone
  Arms: Treatment Group C

SUMMARY:
This study will be conducted to determine the preliminary efficacy of axatilimab in combination with ruxolitinib and to assess the contribution of axatilimab to the combination treatment effect in participants with cGVHD.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 12 years of age at the time of informed consent.
* New-onset moderate or severe cGVHD, as defined by the 2014 NIH Consensus Development Project Criteria for Clinical Trials in cGVHD, requiring systemic therapy.
* History of 1 allo-SCT (any type of stem cell donor, any conditioning regimen, and source of hematopoietic stem cells).
* Adequate hematologic function independent of platelet transfusion and growth factors for at least 7 days prior to study entry: ANC ≥ 0.75 × 109/L and platelet count ≥ 20 × 109/L.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Received more than 1 prior allo-SCT. Prior autologous HCT is allowed.
* Has overlap cGVHD, defined as simultaneous presence of features or characteristics of aGVHD in a patient with cGVHD.
* Received previous systemic treatment for cGVHD, including systemic corticosteroids and extracorporeal photopheresis.
* Received systemic corticosteroids within 2 weeks prior to C1D1, regardless of indication.
* Initiated systemic treatment with CNIs or mTOR inhibitors within 2 weeks prior to C1D1.
* Prior treatment with a JAK inhibitor within 8 weeks before randomization. Participants who received a JAK inhibitor for the treatment of aGVHD are eligible only if they achieved a response (CR or PR) to JAK inhibitor treatment and did not discontinue due to toxicity.
* Evidence of relapse of the primary hematologic disease or treatment for relapse after the allo-SCT was performed, including DLIs for the treatment of molecular relapse.
* History of acute or chronic pancreatitis.
* History of thromboembolic events (such as deep vein thrombosis, pulmonary embolism, stroke, myocardial infarction) in the 6 months prior to study entry.
* Active symptomatic myositis.
* Severe renal impairment, that is, estimated CrCl < 30 mL/min measured or calculated by Cockcroft-Gault equation in adults and Schwartz formula in pediatric participants, or end-stage renal disease on dialysis. Participants with CrCl of 30 to 59 mL/min on treatment with fluconazole are not eligible.
* Impaired liver function, defined as total bilirubin > 1.5 × ULN and/or ALT and AST > 3 × ULN in participants with no evidence of liver cGVHD.
* Currently active significant cardiac disease, such as uncontrolled arrhythmias, uncontrolled hypertension, or Class 3 or 4 congestive heart failure as defined by New York Heart Association, or a history of myocardial infarction or unstable angina within 6 months prior to randomization.
* Pregnant or breastfeeding.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 6 months
  Defined as Complete Response (CR) or Partial Response (PR) at 6 months in the absence of new systemic therapy for cGVHD. Response assessment will be based on the 2014 NIH Consensus Development Project on Criteria for Clinical Trials in cGVHD.

SECONDARY OUTCOMES:
Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to 2 years and 30 days
  Defined as adverse events reported for the first time or worsening of a pre-existing event after the first dose of study treatment.
Duration of Response | Up to 2 years
  Defined as the time from the first response (PR or CR) to the date of progression of cGVHD, start of new systemic therapy or death from any cause.
Proportion of participants with a ≥ 7-point improvement in modified Lee symptom scale (mLSS) score | Up to 2 years
Best overall response in the first 6 months | Up to 6 months
  Define as PR or CR in the first 6 months.
OR at 12 months, defined as CR or PR at 12 months (C14D1) in the absence of new systemic therapy for cGVHD. | 12 months
  Defined as CR or PR at 12 months in the absence of new systemic therapy for cGVHD
Proportion of participants who remain corticosteroid-free | 4 weeks, 8 weeks and 6 months
Organ-specific response in the first 6 cycles and on study, based on the 2014 NIH Consensus Development Project on Criteria for Clinical Trials in cGVHD. | Up to 2 years
  Based on the 2014 NIH Consensus Development Project on Criteria for Clinical Trials in cGVHD.
Failure-free Survival (FFS) | Up to 2 years and 30 days
  Defined as the time from date of randomization to date of initiation of a new cGVHD treatment, malignancy relapse, or death due to any cause.
Axatilimab pharmacokinetic (PK) in Plasma | Up to 2 years and 30 days
  Axatilimab concentration in plasma.
Ruxolitinib PK in Plasma | Up to 2 years and 30 days
  Ruxolitinib concentration in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (70):
- United States (26):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - City of Hope Medical Center, Duarte, California
  - University of California-Los Angeles Medl Cntr-Oncology Center Bowyer Clinic, Los Angeles, California
  - Stanford Cancer Center, Stanford, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Smilow Cancer Center-Yale, New Haven, Connecticut
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - The University of Chicago Medicine, Chicago, Illinois
  - University of Maryland-Greenebaum Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Fred and Pamela Buffett Cancer Center, Omaha, Nebraska
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Md Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington, Seattle, Washington
  - Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin
- Belgium (7):
  - Az Sint-Jan Brugge - Oostende Av - Campus Sint-Jan, Bruges
  - Universitair Ziekenhuis Antwerpen (Uza), Edegem
  - Jessa Ziekenhuis, Hasselt
  - Universitair Ziekenhuis (Uz) Leuven, Leuven
  - Universitaire Ziekenhuis Leuven - Gasthuisberg, Leuven
  - Centre Hospitalier Universitaire (Chu) de Liege, Liège
  - AZ DELTA, Roeselare
- Canada (4):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Princess Margaret Cancer Centre - University Health Network, Toronto, Ontario
  - Chu Sainte-Justine, Montreal, Quebec
  - Vancouver General Hospital, Vancouver
- Germany (6):
  - Klinikum Der Johann Wolfgang Goethe University, Frankfurt am Main
  - Universitatklinikum Freiburg, Freiburg im Breisgau
  - Universitatsklinikum Hamburg Eppendorf, Hamburg
  - Universitaetsklinikum Jena, Jena
  - University Hospital Mannheim, Mannheim
  - Universitaetsklinikum Regensburg, Regensburg
- Italy (7):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni Xxiii, Bergamo
  - Aou Policlinico S. Orsola-Malpighi, Bologna
  - Fondazione Irccs Ca Granda Ospedale Maggiore Policlinico Di Milano Uo Dermatologia, Milan
  - Ospedale Pediatrico Bambino Gesu Irccs, Rome
  - Policlinico Universitario Agostino Gemelli Universita Cattolica Del Sacro Cuore, Rome
  - Irccs Istituto Clinico Humanitas, Rozzano
  - A.O.U. Citta Della Salute E Della Scienza Di Torino, Torino
- Spain (14):
  - Hospital General Universitario Vall D Hebron, Barcelona
  - Hospital Clinic Barcelona Main, Barcelona
  - Hospital Universitario Virgen de La Arrixaca, El Palmar
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Ico Institut Catala D Oncologia, Granvia de L'hospitalet 199-203
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitari I Politecnic La Fe, Valencia
- United Kingdom (6):
  - Queen Elizabeth Hospital, Birmingham
  - Cambridge University Hospitals Nhs Foundation Trust, Cambridge
  - University Hospital of Wales, Cardiff
  - Queen Elizabeth University Hospital, Glasgow
  - St James University Hospital, Leeds
  - Clatterbridge Cancer Center, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: A Study to Evaluate the Safety and Efficacy of Axatilimab in Combination With Ruxolitinib in Participants With Newly Diagnosed Chronic Graft-Versus-Host Disease — https://www.incyteclinicaltrials.com/study/?id=INCA34176-254&SearchTerm=INCA34176-254&Latitude=&Longitude=&LocationName=&conditions=&Status=&phases=&AgeRanges=&gender=&StudyTypes=&AttachmentTypes=&MileRadius=100&PageIndex=0&PageSize=10&SortField=&SortOrder=&hasResults=